CLINICAL TRIAL: NCT01518114
Title: Exercise Training in Patients With Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Michael Arad, MD, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-10-8081-MA-CTIL
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic Cardiomyopathy; Exercise Training; Cardiac Rehabilitation; Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Heart Failure | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Training (Experimental): Exercise will be performed under continuous telemetry monitoring and medical supervision. Each session will include 5-10 worm-up, 30 min of aerobic activity on treadmill or bicycle ergometer followed by 10-15 min of stretch and relaxation exercise. Blood pressure will be obtained before the onset and at the end of each session. Participants will be requested to rest and observed 15-30 min before going home. The exercise intensity will be monitored and adjusted, per protocol, according to RPE using the Borg scale.
  Exercise prescription will be based upon cardiopulmonary test done at baseline.
  Interventions: Behavioral: Exercise Training
- Best Medical Care (Active Comparator): Advanced HCM patients who are eligible to participate in the study but cannot do so for technical reasons will be invited to participate in the project as a control group.These subjects will continue their regular follow up in the Cardiomyopathy Clinic and their usual voluntary physical activity at home.
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training — Exercise will be performed under continuous telemetry monitoring and medical supervision. Each session will include 5-10 worm-up, 30 min of aerobic activity on treadmill or bicycle ergometer followed by 10-15 min of stretch and relaxation exercise. Blood pressure will be obtained before the onset and at the end of each session. Participants will be requested to rest and observed 15-30 min before going home. The exercise intensity will be monitored and adjusted, per protocol, according to RPE using the Borg scale.

SUMMARY:
Exercise training (ET) is highly beneficial in heart failure patients and has been suggested to confer significant symptomatic and functional improvements in patients with diastolic dysfunction. Accordingly, the aim of this study was to examine the safety, feasibility of a structured ET program in symptomatic HCM patients.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic Cardiomyopathy
* NYHA 3
* Maximal left ventricular wall thickness > 20 mm
* Age >18

Exclusion Criteria:

* Severe non-cardiac limitations of functional capacity such as neurological illness, lung disease, peripheral vascular or orthopedic problem, etc.
* Patients state post resuscitation for malignant ventricular arrhythmia.
* History of effort induced syncope, complex ventricular arrhythmia or atrial fibrillation.
* An exercise-induced decrease in blood pressure
* Severe left ventricular outflow obstruction defined as resting outflow gradient > 50 mmHg on maximal therapy
* Atrial fibrillation with a poorly controlled ventricular response
* Advanced hypokinetic stage of HCM defined as LVEF < 40%
* Congestive heart failure of angina FC IV according to NYHA or CCS respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Functional capacity improvement as determined by the degree of percent change in VO2 MAX following structured exercise rehabilitation | 6 months
  End point to be assessed by cardiopulmonary testing are pre- and post exercise training improvement as expressed by the changes in : VO2 MAX, exercise duration, duration to ventilatory threshold(VT).
Safety of exercise training in patients with symptomatic hypertrophic cardiomyopathy | 12 months
  Safety endpoonts: 1) Clinicaly significant arrhythmia during exercise training 2)MACE during follow-up period (ACS, Stroke or Death) 3)Exercise Related Injury 4) Episodes of syncope

SECONDARY OUTCOMES:
Secondary Endpoints: | 12 months
  1. The effect on quality of life
  2. The change in maximal wall thickness, LVEF, resting and exercise-induced left ventricular outflow gradient and pulmonary artery pressure (stress echo).
  3. Resting BNP and troponin I levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Hashomer , Ramat Gan, Israel